CLINICAL TRIAL: NCT01131351
Title: A Phase 2, Multi-center, Non-controlled, Open-label Dose Escalation Trial to Assess the Safety, Tolerability, Pharmacokinetics, and Efficacy of Orally Administered OPC-67683 Two Times Daily to Patients With Pulmonary Multidrug-Resistant Tuberculosis Refractory to Conventional Treatment
Brief Title: Safety and Pharmacokinetics (PK) in Multidrug-Resistant (MDR) Refractive Tuberculosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated early due to lack of efficacy after 10 participants enrolled.
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 242-08-210; 2009-014944-13 (EudraCT Number)
Record Dates: First submitted 2010-05-25; First posted 2010-05-26 (Estimated); Results first posted 2021-11-11 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-10

CONDITIONS: Tuberculosis
Keywords: MDR-TB; Dose Escalation; Phase II; Open Label; Non Controlled; Pulmonary Multidrug-Resistant Tuberculosis (MDR TB)
MeSH Terms: conditions — Tuberculosis; Tuberculosis, Multidrug-Resistant | interventions — OPC-67683

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Delamanid 250 mg BID+ OBR (Experimental): Participants received delamanid five 50 milligrams (mg) (250 mg) tablets, twice a day (BID), along with at least 2 additional anti-TB medications per optimized background regimen (OBR) for up to 28 weeks.
  Interventions: Drug: Delamanid; Drug: Optimized Background Regimen (OBR)
- Delamanid 300 mg BID+ OBR (Experimental): Participants received delamanid six 50 mg (300 mg) tablets, BID, along with at least 2 additional anti-TB medications per OBR for up to 28 weeks.
  Interventions: Drug: Delamanid; Drug: Optimized Background Regimen (OBR)

INTERVENTIONS:
Drug: Delamanid — OPC-67683 film-coated tablets
  Other Names: OPC-67683
Drug: Optimized Background Regimen (OBR) — OBR was selected at the discretion of the study investigator and included at least 2 anti-TB medications based on World Health Organization (WHO's) guidelines for the programmatic management of drug-resistant TB. Study investigator could change OBR for a participant based on his/her tolerability and drug susceptibility testing (DST) results.

SUMMARY:
The purpose of this study is:

* To evaluate the safety and tolerability of orally administered OPC-67683 when administered two times daily to MDR tuberculosis (TB) participants refractory to treatment with an optimized background regimen of anti-TB medications (OBR).
* To evaluate the pharmacokinetics (PK) of OPC-67683 and metabolites.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written, informed consent prior to all trial-related procedures
2. Male or female participants aged between 18 and 64 years, inclusive.
3. Able to produce sputum for mycobacterium culture or able to obtain sputum produced through Induction.
4. At least three sputum mycobacterium cultures positive for MTB with in-vitro resistance to isoniazid and rifampicin during the previous 270 days (9 months) despite treatment with first and second line anti-TB drugs, including one positive culture within the previous 60 days from the time of sputum collection, prior to date of screening initiation [defined as the date the informed consent form (ICF) is signed and screening begins].
5. Sputum mycobacterial culture positive for MTB with in-vitro susceptibility to at least one anti-TB medication within the previous 60 days prior to the date of screening initiation.
6. Participant judged by the investigator to have potential for clinical benefit from OPC-67683 exposure.
7. Female participants of childbearing potential must have a negative urine pregnancy test and agree to use a highly effective method of birth control (for example, two of the following precautions: tubal ligation, vaginal diaphragm, intrauterine device, oral contraceptives, contraceptive implant, combined hormonal patch, combined injectable contraceptive or depot-medroxyprogesterone acetate) throughout the participation in the trial and for 22 weeks after last dose (to cover duration of ovulation).
8. Male participant must agree to use an adequate method of contraception (double barrier) throughout the participation in the trial and for 30 weeks after last dose (to cover duration of spermatogenesis).

Exclusion Criteria:

1. A history of allergy to any nitro-imidazoles or nitro-imidazole derivatives at any time.
2. Use of the medications in Section 4.1 including: use of amiodarone at any time during the previous 12 months, use of other antiarrhythmics for the previous 30 days, as well as use of certain antidepressants, anti-histamines, any macrolides, for the previous 14 days.
3. Any current serious concomitant conditions or renal impairment characterized by serum creatinine levels ~265 micromoles (μmol)/L or hepatic impairment characterized by alanine aminotransferase (ALT) and/or aspartate transferase (AST) levels 3 times the upper limit of the laboratory reference range.
4. Current clinically relevant changes in the Screening electrocardiogram (ECG) such as any atrioventricular (AV) block, prolongation of the QRS complex over 120 msec (in both male and female participants), or of the QT interval with Fridericia's correction (QTcF) interval over 450 msec in male participants and over 470 msec in female participants.
5. Current clinically relevant cardiovascular disorder such as heart failure, coronary heart disease, uncontrolled or poorly controlled hypertension, arrhythmia, tachyarrhythmia or status after myocardial infarction.
6. For participants with human immunodeficiency virus (HIV) infection, helper/inducer T-lymphocyte (CD4 cell) count < 350/mm^3 or on treatment with anti-retroviral medication for HIV infection.
7. Karnofsky score < 50%.
8. Any current diseases or conditions in which the use of nitro-imidazoles or nitro-imidazole derivates is contra-indicated.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2010-02-19 (Actual); Primary Completion 2011-05-12 (Actual); Study Completion 2011-05-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Infectology Center of Latvia - Clinic of Tuberculosis and Lung Diseases, Ogre, Latvia
- Lithuania (2):
  - Hospital for Tuberculosis and Lung Diseases, Šiauliai
  - National Tuberculosis and Infectious Diseases University Hospital, Vilnius

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims prespecified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on the Vivli data sharing platform which can be found here: https://vivli.org/ourmember/Otsuka/
URL: https://clinical-trials.otsuka.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 3 investigative sites in Latvia and Lithuania from 19 February 2010 to 12 May 2011.
Pre-assignment Details: A total of 10 participants received at least one dose of delamanid (5 participants in delamanid 250 mg BID+ OBR group and 5 participants in delamanid 300 mg BID+ OBR group). Of which, 7 participants completed the study.
Groups:
- Delamanid 250 mg BID + OBR: Participants received delamanid five 50 milligrams (mg) (250 mg) tablets, twice a day (BID), along with at least 2 additional anti-TB medications per optimized background regimen (OBR) for up to 28 weeks.
- Delamanid 300 mg BID + OBR: Participants received delamanid six 50 mg (300 mg) tablets, BID, along with at least 2 additional anti-TB medications per OBR for up to 28 weeks.
Period: Overall Study
Arm/Group | Delamanid 250 mg BID + OBR | Delamanid 300 mg BID + OBR
Started | 5 | 5
Completed | 5 | 2
Not Completed | 0 | 3
Not completed — Adverse Event | 0 | 2
Not completed — Protocol Deviation | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) Population included all participants who took at least one dose of investigational medicinal product (IMP).
Groups:
- Delamanid 250 mg BID + OBR: Participants received delamanid five 50 mg (250 mg) tablets, BID, along with at least 2 additional anti-TB medications per OBR for up to 28 weeks.
- Total: Total of all reporting groups
Arm/Group | Delamanid 250 mg BID + OBR | Delamanid 300 mg BID + OBR | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.6 (10.8) | 34.0 (12.5) | 40.3 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 5 | 4 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 5 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 5 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Potentially Clinically Significant Abnormalities in Vital Signs
Description: Vital signs included body weight [kilogram (kg)], body temperature [degree Celsius (°C)], heart rate [beats per minute (BPM)], respiratory rate (breaths/minute), systolic and diastolic blood pressure [millimeter of mercury (mmHg)]. The criteria for clinically significant abnormal value were: body weight (kg): increase >=5% or decrease >=5%; body temperature (°C): >=38.5°C and increase of >=1.1°C; heart rate (BPM): >=120 bpm and increase of >=15 bpm, or <=60 bpm and decrease of >=15 bpm; systolic blood pressure (mmHg): >=160 mmHg and increase of >=20 mmHg, or <=90 mmHg and decrease of >=20 mmHg; diastolic blood pressure (mmHg): >=105 mmHg and increase of >=15 mmHg, or <=50 mmHg and decrease of >=15 mmHg; respiration rate (breaths per minute) >30 breaths per minute. Only categories with data for potentially clinically significant abnormal vital sign parameter values are reported.
Time Frame: Up to approximately 40 weeks
Population: Safety Analysis Population included all participants who received at least one dose (partial dose inclusive) of trial medication. Number analyzed is the number of participants who had at least one post-baseline numerical result for the given test. Baseline was defined as the last measurements prior to the first dosing of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Delamanid 250 mg BID + OBR | Delamanid 300 mg BID + OBR
Number analyzed (Participants) | 5 | 5
percentage of participants
  Weight: Decrease of >=5% in Body Weight | 60.0 | 0.0
  Weight: Increase of >=5% in Body Weight | 20.0 | 0.0
  Heart Rate: <=60 bpm + Decrease of >=15 bpm | 40.0 | 20.0
  Systolic Blood Pressure: <= 90 mmHg + Decrease of >=20 mmHg | 40.0 | 0.0
  Respiration Rate: >30 Breaths Per Minute | 20.0 | 0.0

2. Primary Outcome: Percentage of Participants With Potentially Clinically Significant Abnormalities in Electrocardiogram (ECG) Results
Description: The criteria for clinically significant abnormal ECG values were- ventricular rate outlier (<50 bpm and decrease of >=25%, >100 bpm and increase of >=25%), PR outlier [increase of >=25% when PR >200 milliseconds (ms)], QRS outlier (increase of >=25% when QRS >100 ms), QT (new onset (in treatment period but not at Baseline) [>500 ms]), QT interval corrected by Bazett's formula (QTcB) (new onset [>450, >480, >500 ms], increase of >=30 ms and <= 60 ms or increase of >60 ms), QT interval corrected by Fridericia's formula (QTcF) (new onset [>450, >480, >500 ms], increase of >=30 ms and <= 60 ms or increase of >60 ms), new abnormal U waves, new ST segment changes, new T wave changes, new abnormal rhythm, new conduction abnormality were reported as categories. Baseline was defined as the average of the ECGs taken at Day -1. Only categories with data for potentially clinically significant abnormal ECG values are reported.
Time Frame: Up to approximately 40 weeks
Population: Safety Analysis Population included all participants who received at least one dose (partial dose inclusive) of trial medication.
Measure: Number; unit: percentage of participants
Arm/Group | Delamanid 250 mg BID + OBR | Delamanid 300 mg BID + OBR
Number analyzed (Participants) | 5 | 5
percentage of participants
  Vent Rate Outliers: Notable Decreases | 40.00 | 0.00
  Vent Rate Outliers: Notable Increases | 40.00 | 0.00
  QTcB: New Onset (>500 msec) | 0.00 | 20.00
  QTcB: New Onset (>480 msec) | 0.00 | 40.00
  QTcB: New Onset (>450 msec) | 40.00 | 40.00
  QTcB: Change >=30, <=60 msec | 40.00 | 80.00
  QTcF: New Onset (>500 msec) | 0.00 | 20.00
  QTcF: New Onset (>480 msec) | 0.00 | 20.00
  QTcF: New Onset (>450 msec) | 0.00 | 40.00
  QTcF: Change >=30, <=60 msec | 60.00 | 80.00
  ST Segment: New ST Segment Changes | 0.00 | 20.00
  T Waves: New T Wave Changes | 20.00 | 20.00
  Rhythm: New Abnormal Rhythm | 60.00 | 80.00
  Conduction: New Conduction Changes | 0.00 | 40.00

3. Primary Outcome: Percentage of Participants With Potentially Clinically Significant Laboratory Values
Description: Clinical laboratory tests included hematology, coagulation, chemistry, and urinalysis. The participants were categorized based on the clinically significant laboratory values as per protocol predefined criteria. The categories with at least one participant with clinically significant value outside the normal range for laboratory assessments are reported.
Time Frame: Up to approximately 40 weeks
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Delamanid 250 mg BID + OBR | Delamanid 300 mg BID + OBR
Number analyzed (Participants) | 5 | 5
percentage of participants
  Lactic Dehydrogenase [units per liter (U/L)] | 0.0 | 20.0
  Potassium [milliequivalents per liter (mEq/L)] | 60.0 | 20.0
  Sodium (mEq/L) | 0.0 | 20.0
  Triglycerides [milligrams per deciliter (mg/dL)] | 0.0 | 20.0
  Uric acid (mg/dL) | 0.0 | 20.0
  Lymphocytes [percentage (%)] | 0.0 | 20.0
  Lymphocytes, Absolute [thousand cells per microliter (thous/µL)] | 0.0 | 20.0
  Mean Corpuscular Volume [femtoliter (fL)] | 20.0 | 20.0
  Neutrophils, Absolute (thous/µL) | 0.0 | 20.0
  Platelet Count (thous/µL) | 20.0 | 0.0
  Prothrombin Time [seconds (sec)] | 0.0 | 20.0
  Red Blood Cell Count [million cells per microliter (mill/µL)] | 20.0 | 20.0
  Reticulocyte Count (%) | 60.0 | 60.0

4. Primary Outcome: Percentage of Participants With Abnormal Audiometry Assessment Values
Time Frame: Up to approximately 40 weeks
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Delamanid 250 mg BID + OBR | Delamanid 300 mg BID + OBR
Number analyzed (Participants) | 5 | 5
percentage of participants | 100.0 | 80.0

5. Primary Outcome: Percentage of Participants With Abnormal Visual Acuity Assessment Values
Time Frame: Up to approximately 40 weeks
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Delamanid 250 mg BID + OBR | Delamanid 300 mg BID + OBR
Number analyzed (Participants) | 5 | 5
percentage of participants | 40.0 | 20.0

6. Primary Outcome: Percentage of Participants Taking Concomitant Anti-Tuberculosis (TB) Medication During the Trial
Time Frame: Up to approximately 40 weeks
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Delamanid 250 mg BID + OBR | Delamanid 300 mg BID + OBR
Number analyzed (Participants) | 5 | 5
percentage of participants
  Total Participants Using One or More Medications | 100.0 | 100.0
  Participants Taking Antibacterials for Systemic Use | 80.0 | 80.0
  Participants Taking Antimycobacterials | 100.0 | 100.0

7. Primary Outcome: Percentage of Participants Taking Concomitant (Excluding Anti-TB) Medication During the Trial
Time Frame: Up to approximately 40 weeks
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Delamanid 250 mg BID + OBR | Delamanid 300 mg BID + OBR
Number analyzed (Participants) | 5 | 5
percentage of participants
  Total Participants Using One or More Medications | 100.0 | 100.0
  Participants Taking Agents Acting on the Renin-Angiotensin System | 20.0 | 20.0
  Participants Taking Analgesics | 40.0 | 0.0
  Participants Taking Antidiarrheals, Intestinal Antiinflammatory | 20.0 | 0.0
  Participants Taking Antiepileptics | 20.0 | 0.0
  Participants Taking Antigout Preparations | 0.0 | 20.0
  Participants Taking Antihemorrhagics | 20.0 | 20.0
  Participants Taking Antihypertensives | 20.0 | 0.0
  Participants Taking Antiinflammatory and Antirheumatic Products | 60.0 | 20.0
  Participants Taking Antimycotics for Systemic Use | 0.0 | 20.0
  Participants Taking Blood Substitutes and Perfusion Solutions | 40.0 | 40.0
  Participants Taking Cardiac Therapy | 0.0 | 20.0
  Participants Taking Corticosteroids for Systemic Use | 0.0 | 40.0
  Participants Taking Cough and Cold Preparations | 60.0 | 40.0
  Participants Taking Digestives, Including Enzymes | 80.0 | 20.0
  Participants Taking Diuretics | 40.0 | 0.0
  Participants Taking Drugs for Acid Related Disorders | 80.0 | 40.0
  Participants Taking Drugs for Functional Gastrointestinal Disorders | 60.0 | 0.0
  Participants Taking Drugs for Obstructive Airway Diseases | 40.0 | 100.0
  Participants Taking Nasal Preparations | 0.0 | 20.0
  Participants Taking Otologicals | 0.0 | 20.0
  Participants Taking Psycholeptics | 60.0 | 40.0
  Participants Taking Unspecified Herbal and Traditional Medicine | 40.0 | 100.0
  Participants Taking Vasoprotectives | 20.0 | 0.0
  Participants Taking Vitamins | 0.0 | 60.0

8. Primary Outcome: Percentage of Participants With Adverse Events (AEs)
Description: An AE was defined as any new medical problem, or exacerbation of an existing problem, experienced by a participant while enrolled in the trial, whether or not it was considered drug-related by the investigator.
Time Frame: Up to approximately 40 weeks
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Delamanid 250 mg BID + OBR | Delamanid 300 mg BID + OBR
Number analyzed (Participants) | 5 | 5
percentage of participants | 100.0 | 100.0

9. Primary Outcome: Percentage of Participants With Immediately Reportable Events (IREs)
Description: An AE was considered serious if it was fatal; life-threatening; persistently or significantly disabling or incapacitating; required in-participant hospitalization or prolonged hospitalization; a congenital anomaly/birth defect; or other medically significant event that, based upon appropriate medical judgment, may have jeopardized the participant and may have required medical or surgical intervention to prevent one of the outcomes listed above. The following were considered as IREs- serious adverse events (SAEs), pregnancies in trial participants or their partners, and all events involving overdose, misuse and abuse.
Time Frame: Up to approximately 40 weeks
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Delamanid 250 mg BID + OBR | Delamanid 300 mg BID + OBR
Number analyzed (Participants) | 5 | 5
percentage of participants | 40.0 | 40.0

10. Primary Outcome: Cmax: Maximal Peak Plasma Concentration for Delamanid
Time Frame: At 24 hours post dose on Days 1, 14, 28, 56, 112 and 196
Population: Intent-to-treat (ITT) Population included all participants who took at least one dose of IMP. Number analyzed is the number of participants with evaluable data at the given time point.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Delamanid 250 mg BID + OBR | Delamanid 300 mg BID + OBR
Number analyzed (Participants) | 5 | 5
nanograms per milliliter (ng/mL)
  Day 1 | 142 (68.2) | 192 (93.5)
  Day 14 | 521 (132) | 514 (99.3)
  Day 28 | 558 (113) | 573 (117)
  Day 56 | 558 (239) | 503 (126)
  Day 112: number analyzed (Participants) | 5 | 4
  Day 112 | 441 (286) | 427 (114)
  Day 196: number analyzed (Participants) | 5 | 2
  Day 196 | 494 (129) | 499 (241)

11. Primary Outcome: Tmax: Time to Reach Maximal Peak Plasma Concentration for Delamanid
Time Frame: At 24 hours post dose on Days 1, 14, 28, 56, 112 and 196
Population: ITT Population included all participants who took at least one dose of IMP. Number analyzed is the number of participants with evaluable data at the given time point.
Measure: Median (Full Range); unit: hours
Arm/Group | Delamanid 250 mg BID + OBR | Delamanid 300 mg BID + OBR
Number analyzed (Participants) | 5 | 5
hours
  Day 1 | 2.95 [2.95 to 12.15] | 3.20 [3.00 to 11.88]
  Day 14 | 2.95 [0.00 to 3.27] | 3.02 [2.53 to 3.05]
  Day 28 | 2.95 [2.95 to 3.00] | 3.03 [3.00 to 8.92]
  Day 56 | 2.95 [0.00 to 8.95] | 3.00 [3.00 to 8.97]
  Day 112: number analyzed (Participants) | 5 | 4
  Day 112 | 2.95 [0.00 to 3.00] | 3.03 [3.00 to 3.05]
  Day 196: number analyzed (Participants) | 5 | 2
  Day 196 | 2.95 [0.00 to 8.95] | 3.00 [3.00 to 3.00]

12. Primary Outcome: AUC0-24h: Area Under the Plasma Concentration-Time Curve From 0 To 24 Hours for Delamanid
Description: AUC0-24h was calculated as 2×AUC0-12h.
Time Frame: At 24 hours post dose on Days 1, 14, 28, 56, 112 and 196
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: hour*nanograms per milliliter (h*ng/mL)
Arm/Group | Delamanid 250 mg BID + OBR | Delamanid 300 mg BID + OBR
Number analyzed (Participants) | 5 | 5
hour*nanograms per milliliter (h*ng/mL)
  Day 1 | 2020 (708) | 2650 (1280)
  Day 14 | 9580 (2790) | 10400 (1950)
  Day 28 | 9840 (3090) | 11200 (2450)
  Day 56 | 10500 (4490) | 9720 (2400)
  Day 112: number analyzed (Participants) | 5 | 4
  Day 112 | 8020 (5470) | 8470 (3080)
  Day 196: number analyzed (Participants) | 5 | 2
  Day 196 | 9420 (2340) | 8640 (2890)

13. Primary Outcome: Rac (Cmax): Ratio of Accumulation for Cmax of Delamanid
Description: Ratio of accumulation for Cmax was assessed on Days 14, 28, 56, 112 and 196 with respect to Day 1.
Time Frame: At 24 hours post dose on Days 1, 14, 28, 56, 112 and 196
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Delamanid 250 mg BID + OBR | Delamanid 300 mg BID + OBR
Number analyzed (Participants) | 5 | 5
ratio
  Day 1: number analyzed (Participants) | 0 | 0
  Day 14 | 4.01 (1.22) | 3.76 (3.13)
  Day 28 | 4.33 (1.31) | 4.01 (2.84)
  Day 56 | 4.04 (0.657) | 3.24 (1.71)
  Day 112: number analyzed (Participants) | 5 | 4
  Day 112 | 3.07 (1.25) | 1.89 (0.485)
  Day 196: number analyzed (Participants) | 5 | 2
  Day 196 | 3.80 (1.25) | 1.93 (0.418)

14. Primary Outcome: Rac (AUC): Ratio of Accumulation for AUC of Delamanid
Description: Ratio of accumulation for AUC was assessed on Days 14, 28, 56, 112 and 196 with respect to Day 1.
Time Frame: At 24 hours post dose on Days 1, 14, 28, 56, 112 and 196
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Delamanid 250 mg BID + OBR | Delamanid 300 mg BID + OBR
Number analyzed (Participants) | 5 | 5
ratio
  Day 1: number analyzed (Participants) | 0 | 0
  Day 14 | 4.85 (0.938) | 5.45 (4.38)
  Day 28 | 4.92 (0.699) | 5.66 (4.18)
  Day 56 | 5.13 (0.762) | 4.55 (2.45)
  Day 112: number analyzed (Participants) | 5 | 4
  Day 112 | 3.74 (1.47) | 2.85 (1.27)
  Day 196: number analyzed (Participants) | 5 | 2
  Day 196 | 4.79 (0.800) | 2.29 (0.367)

15. Secondary Outcome: Cmax: Maximal Peak Plasma Concentration for Delamanid Metabolites
Description: The primary metabolites of delamanid are DM-6704, DM-6705 and DM-6706.
Time Frame: At 24 hours post dose on Days 1, 14, 28, 56, 112 and 196
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Delamanid 250 mg BID + OBR | Delamanid 300 mg BID + OBR
Number analyzed (Participants) | 5 | 5
ng/mL
  DM-6704: Cmax at Day 1: number analyzed (Participants) | 3 | 3
  DM-6704: Cmax at Day 1 | 1.33 (0.257) | 2.53 (1.59)
  DM-6704: Cmax at Day 14 | 43.1 (25.2) | 82.7 (32.8)
  DM-6704: Cmax at Day 28 | 52.5 (12.8) | 95.9 (31.5)
  DM-6704: Cmax at Day 56 | 59.9 (22.4) | 119 (79.6)
  DM-6704: Cmax at Day 112: number analyzed (Participants) | 5 | 4
  DM-6704: Cmax at Day 112 | 58.5 (33.8) | 88.8 (67.3)
  DM-6704: Cmax at Day 196: number analyzed (Participants) | 5 | 2
  DM-6704: Cmax at Day 196 | 71.2 (8.85) | 99.3 (104)
  DM-6705: Cmax at Day 1 | 2.88 (1.41) | 3.75 (1.79)
  DM-6705: Cmax at Day 14 | 76.6 (25.4) | 95.4 (30.1)
  DM-6705: Cmax at Day 28 | 114 (47.8) | 146 (58.8)
  DM-6705: Cmax at Day 56 | 140 (64.2) | 142 (50.1)
  DM-6705: Cmax at Day 112: number analyzed (Participants) | 5 | 4
  DM-6705: Cmax at Day 112 | 128 (85.0) | 126 (80.2)
  DM-6705: Cmax at Day 196: number analyzed (Participants) | 5 | 2
  DM-6705: Cmax at Day 196 | 135 (62.9) | 154 (128)
  DM-6706: Cmax at Day 1: number analyzed (Participants) | 0 | 0
  DM-6706: Cmax at Day 14 | 44.6 (24.1) | 71.9 (23.1)
  DM-6706: Cmax at Day 28 | 64.0 (27.9) | 97.7 (23.0)
  DM-6706: Cmax at Day 56 | 77.6 (28.4) | 103 (72.2)
  DM-6706: Cmax at Day 112: number analyzed (Participants) | 5 | 4
  DM-6706: Cmax at Day 112 | 75.2 (36.5) | 83.1 (54.7)
  DM-6706: Cmax at Day 196: number analyzed (Participants) | 5 | 2
  DM-6706: Cmax at Day 196 | 81.7 (6.38) | 94.9 (92.1)

16. Secondary Outcome: Tmax: Time to Reach Maximal Peak Plasma Concentration for Delamanid Metabolites
Description: The primary metabolites of delamanid are DM-6704, DM-6705 and DM-6706.
Time Frame: At 24 hours post dose on Days 1, 14, 28, 56, 112 and 196
Population: as for outcome 11
Measure: Median (Full Range); unit: hours
Arm/Group | Delamanid 250 mg BID + OBR | Delamanid 300 mg BID + OBR
Number analyzed (Participants) | 5 | 5
hours
  DM-6704: Tmax at Day 1: number analyzed (Participants) | 3 | 3
  DM-6704: Tmax at Day 1 | 11.95 [8.95 to 12.15] | 12.00 [11.88 to 12.25]
  DM-6704: Tmax at Day 14 | 2.95 [0.00 to 12.12] | 3.02 [0.00 to 12.00]
  DM-6704: Tmax at Day 28 | 2.95 [0.00 to 2.95] | 3.00 [0.00 to 8.92]
  DM-6704: Tmax at Day 56 | 5.95 [0.00 to 8.95] | 3.00 [0.00 to 9.00]
  DM-6704: Tmax at Day 112: number analyzed (Participants) | 5 | 4
  DM-6704: Tmax at Day 112 | 0.00 [0.00 to 11.95] | 0.00 [0.00 to 9.00]
  DM-6704: Tmax at Day 196: number analyzed (Participants) | 5 | 2
  DM-6704: Tmax at Day 196 | 2.95 [0.00 to 8.95] | 3.00 [3.00 to 3.00]
  DM-6705: Tmax at Day 1 | 5.95 [2.95 to 12.15] | 5.92 [3.00 to 12.25]
  DM-6705: Tmax at Day 14 | 5.95 [0.00 to 11.95] | 9.00 [3.02 to 11.53]
  DM-6705: Tmax at Day 28 | 2.95 [2.95 to 5.95] | 6.00 [3.03 to 8.92]
  DM-6705: Tmax at Day 56 | 5.95 [2.95 to 9.00] | 8.97 [0.00 to 12.00]
  DM-6705: Tmax at Day 112: number analyzed (Participants) | 5 | 4
  DM-6705: Tmax at Day 112 | 2.95 [0.00 to 8.95] | 3.00 [0.00 to 6.03]
  DM-6705: Tmax at Day 196: number analyzed (Participants) | 5 | 2
  DM-6705: Tmax at Day 196 | 5.95 [2.95 to 12.00] | 7.49 [6.00 to 8.98]
  DM-6706: Tmax at Day 1: number analyzed (Participants) | 0 | 0
  DM-6706: Tmax at Day 14 | 8.95 [0.00 to 12.12] | 0.00 [0.00 to 5.97]
  DM-6706: Tmax at Day 28 | 2.95 [2.95 to 12.00] | 3.00 [0.00 to 8.92]
  DM-6706: Tmax at Day 56 | 5.95 [0.00 to 8.95] | 0.00 [0.00 to 9.00]
  DM-6706: Tmax at Day 112: number analyzed (Participants) | 5 | 4
  DM-6706: Tmax at Day 112 | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 12.00]
  DM-6706: Tmax at Day 196: number analyzed (Participants) | 5 | 2
  DM-6706: Tmax at Day 196 | 8.95 [2.95 to 8.98] | 6.01 [3.00 to 9.02]

17. Secondary Outcome: AUC0-24h: Area Under the Plasma Concentration-Time Curve From 0 To 24 Hours for Delamanid Metabolites
Description: The primary metabolites of delamanid are DM-6704, DM-6705 and DM-6706.
Time Frame: At 24 hours post dose on Days 1, 14, 28, 56, 112 and 196
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Delamanid 250 mg BID + OBR | Delamanid 300 mg BID + OBR
Number analyzed (Participants) | 5 | 5
h*ng/mL
  DM-6704: AUC0-24h at Day 1: number analyzed (Participants) | 1 | 1
  DM-6704: AUC0-24h at Day 1 | 11.1 (NA) — The standard deviation was not estimable due to fewer number of participants with data available for analysis. | 19.2 (NA) — The standard deviation was not estimable due to fewer number of participants with data available for analysis.
  DM-6704: AUC0-24h at Day 14 | 928 (567) | 1830 (705)
  DM-6704: AUC0-24h at Day 28 | 1140 (357) | 2100 (666)
  DM-6704: AUC0-24h at Day 56 | 1280 (499) | 2610 (1760)
  DM-6704: AUC0-24h at Day 112: number analyzed (Participants) | 5 | 4
  DM-6704: AUC0-24h at Day 112 | 1220 (711) | 1820 (1250)
  DM-6704: AUC0-24h at Day 196: number analyzed (Participants) | 5 | 2
  DM-6704: AUC0-24h at Day 196 | 1550 (176) | 2130 (2230)
  DM-6705: AUC0-24h at Day 1: number analyzed (Participants) | 5 | 4
  DM-6705: AUC0-24h at Day 1 | 45.5 (13.6) | 64.8 (11.5)
  DM-6705: AUC0-24h at Day 14 | 1650 (543) | 2070 (593)
  DM-6705: AUC0-24h at Day 28 | 2500 (1110) | 3140 (1140)
  DM-6705: AUC0-24h at Day 56 | 3100 (1480) | 3150 (1130)
  DM-6705: AUC0-24h at Day 112: number analyzed (Participants) | 5 | 4
  DM-6705: AUC0-24h at Day 112 | 2790 (1800) | 2710 (1500)
  DM-6705: AUC0-24h at Day 196: number analyzed (Participants) | 5 | 2
  DM-6705: AUC0-24h at Day 196 | 3060 (1410) | 3440 (2890)
  DM-6706: AUC0-24h at Day 1: number analyzed (Participants) | 0 | 0
  DM-6706: AUC0-24h at Day 14 | 966 (531) | 1590 (496)
  DM-6706: AUC0-24h at Day 28 | 1430 (668) | 2190 (498)
  DM-6706: AUC0-24h at Day 56 | 1670 (608) | 2290 (1650)
  DM-6706: AUC0-24h at Day 112: number analyzed (Participants) | 5 | 4
  DM-6706: AUC0-24h at Day 112 | 1630 (815) | 1760 (1050)
  DM-6706: AUC0-24h at Day 196: number analyzed (Participants) | 5 | 2
  DM-6706: AUC0-24h at Day 196 | 1820 (188) | 2060 (2060)

18. Secondary Outcome: Rac (Cmax): Ratios of Accumulation for Cmax for Delamanid Metabolites
Description: The primary metabolites of delamanid are DM-6704, DM-6705 and DM-6706. Ratio of accumulation for Cmax was planned to be assessed on Days 14, 28, 56, 112 and 196 with respect to Day 1.
Time Frame: At 24 hours post dose on Days 1, 14, 28, 56, 112 and 196
Population: Due to limited metabolite exposure on Day 1, the Rac for metabolites was not estimated and hence data was not collected for this endpoint.
Arm/Group | Delamanid 250 mg BID + OBR | Delamanid 300 mg BID + OBR
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Rac (AUC): Ratios of Accumulation for AUC for Delamanid Metabolites
Description: The primary metabolites of delamanid are DM-6704, DM-6705 and DM-6706. Ratio of accumulation for AUC was planned to be assessed on Days 14, 28, 56, 112 and 196 with respect to Day 1. Limited metabolite exposure on Day 1 did not allow for estimation of Rac for metabolites.
Time Frame: At 24 hours post dose on Days 1, 14, 28, 56, 112 and 196
Population: as for outcome 18
Arm/Group | Delamanid 250 mg BID + OBR | Delamanid 300 mg BID + OBR
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: Percentage of Participants With Sputum Culture Conversion by Mycobacteria Growth Indicator Tube (MGIT) at Day 168
Description: Sputum culture conversion was evaluated using the MGIT culture system. A participant was classified as demonstrating a sputum culture conversion if he/she achieved two consecutive sputum cultures negative for growth of Mycobacterium tuberculosis at least 28 days apart after his/her last sputum culture positive for growth and not followed by any sputum specimens positive for growth.
Time Frame: Day 168 (Week 24)
Population: ITT Population included all participants who took at least one dose of IMP.
Measure: Number; unit: percentage of participants
Arm/Group | Delamanid 250 mg BID + OBR | Delamanid 300 mg BID + OBR
Number analyzed (Participants) | 5 | 5
percentage of participants | 0.0 | 20.0

21. Secondary Outcome: Percentage of Participants With Sputum Culture Conversion on Solid Mycobacterial Culture Media at Day 168
Description: Sputum culture status was determined using solid mycobacterial culture media and measuring colony counts per milliliter of sputum. The unit for colony counts: log10 colony-forming unit (CFU)/mL. A participant was classified as demonstrating a sputum culture conversion if he/she achieved two consecutive sputum cultures negative for growth of Mycobacterium tuberculosis at least 28 days apart after his/her last sputum culture positive for growth and not followed by any sputum specimens positive for growth.
Time Frame: Day 168 (Week 24)
Population: ITT Population included all participants who took at least one dose of IMP.
Measure: Number; unit: percentage of participants
Arm/Group | Delamanid 250 mg BID + OBR | Delamanid 300 mg BID + OBR
Number analyzed (Participants) | 5 | 5
percentage of participants | 0.0 | 20.0

22. Secondary Outcome: Mean Change From Baseline in Time to Culture Positivity Using MGIT
Description: The value for time to positivity was defined (in days) as the time interval from inoculation until a positive signal was detected for MTB on sputum culture in the MGIT system during the routine 42 day incubation period. Time to positivity analysis was based on the corresponding qualitative sputum results of positive and negative sputum cultures in days of the initial positive signal for a culture from the MGIT system. Mean is reported for Baseline and mean change from baseline is reported for Days 7, 14, 21, 28, 35, 42, 49, 56, 70, 84, 98, 112, 126, 140, 154, 168, 182, 196, 224, 252, and 280. Baseline is Day -2 and -1. Mean time to culture positivity at Baseline was defined as the average of Day -2 and Day -1 values, if the cultures on both days were positive; and if only one culture was positive, the value for the positive culture was used as baseline.
Time Frame: Baseline and Days 7, 14, 21, 28, 35, 42, 49, 56, 70, 84, 98, 112, 126, 140, 154, 168, 182, 196, 224, 252, and 280
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Delamanid 250 mg BID + OBR | Delamanid 300 mg BID + OBR
Number analyzed (Participants) | 5 | 5
days
  Baseline | 7.7 (3.7) | 6.8 (1.6)
  Change from Baseline at Day 7: number analyzed (Participants) | 5 | 4
  Change from Baseline at Day 7 | 6.8 (12.2) | 3.5 (2.9)
  Change from Baseline at Day 14: number analyzed (Participants) | 5 | 4
  Change from Baseline at Day 14 | 0.7 (1.0) | 1.7 (1.4)
  Change from Baseline at Day 21 | 2.6 (0.9) | 2.1 (2.0)
  Change from Baseline at Day 28: number analyzed (Participants) | 5 | 4
  Change from Baseline at Day 28 | 0.9 (2.7) | 2.1 (2.5)
  Change from Baseline at Day 35: number analyzed (Participants) | 5 | 4
  Change from Baseline at Day 35 | 8.8 (11.1) | 11.1 (15.1)
  Change from Baseline at Day 42 | 6.4 (8.7) | 6.3 (9.9)
  Change from Baseline at Day 49: number analyzed (Participants) | 4 | 4
  Change from Baseline at Day 49 | 0.8 (2.6) | 9.1 (16.4)
  Change from Baseline at Day 56 | 7.3 (11.9) | 5.8 (7.6)
  Change from Baseline at Day 70 | 7.7 (11.9) | 16.4 (16.9)
  Change from Baseline at Day 84: number analyzed (Participants) | 4 | 4
  Change from Baseline at Day 84 | 10.5 (12.4) | 12.1 (16.2)
  Change from Baseline at Day 98: number analyzed (Participants) | 4 | 4
  Change from Baseline at Day 98 | 3.4 (3.9) | 9.8 (16.5)
  Change from Baseline at Day 112: number analyzed (Participants) | 4 | 3
  Change from Baseline at Day 112 | 3.8 (7.0) | 10.7 (20.0)
  Change from Baseline at Day 126: number analyzed (Participants) | 4 | 2
  Change from Baseline at Day 126 | -0.8 (2.9) | 0.1 (1.9)
  Change from Baseline at Day 140: number analyzed (Participants) | 3 | 2
  Change from Baseline at Day 140 | 1.5 (5.4) | 17.3 (25.2)
  Change from Baseline at Day 154: number analyzed (Participants) | 2 | 4
  Change from Baseline at Day 154 | 0.8 (2.1) | 8.3 (17.0)
  Change from Baseline at Day 168: number analyzed (Participants) | 3 | 2
  Change from Baseline at Day 168 | -0.8 (4.5) | 17.3 (23.2)
  Change from Baseline at Day 182: number analyzed (Participants) | 4 | 2
  Change from Baseline at Day 182 | -2.5 (3.0) | 16.5 (24.4)
  Change from Baseline at Day 196: number analyzed (Participants) | 5 | 2
  Change from Baseline at Day 196 | -0.6 (3.9) | 20.9 (18.1)
  Change from Baseline at Day 224: number analyzed (Participants) | 5 | 2
  Change from Baseline at Day 224 | 1.6 (4.6) | 16.2 (24.8)
  Change from Baseline at Day 252: number analyzed (Participants) | 5 | 2
  Change from Baseline at Day 252 | 9.1 (12.0) | 16.5 (24.4)
  Change from Baseline at Day 280: number analyzed (Participants) | 5 | 2
  Change from Baseline at Day 280 | 20.3 (19.0) | 16.6 (24.2)

ADVERSE EVENTS:
Time Frame: From first dose of study drug through end of study (Up to approximately 40 weeks)
Description: Safety Analysis Population included all participants who received at least one dose (partial dose inclusive) of trial medication.
Arm/Group | Delamanid 250 mg BID + OBR | Delamanid 300 mg BID + OBR
All-Cause Mortality (participants affected / at risk) | 0/5 | 1/5
Serious Adverse Events (participants affected / at risk) | 2/5 | 2/5
Other Adverse Events (participants affected / at risk) | 5/5 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Delamanid 250 mg BID + OBR (N=5) | Delamanid 300 mg BID + OBR (N=5)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1
Tuberculosis (Infections and infestations) | 0 | 2
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 1
Alcohol abuse (Psychiatric disorders) | 0 | 1
Lung lobectomy (Surgical and medical procedures) | 2 | 0
Pneumonectomy (Surgical and medical procedures) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Delamanid 250 mg BID + OBR (N=5) | Delamanid 300 mg BID + OBR (N=5)
Anaemia (Blood and lymphatic system disorders) | 2 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 3 | 1
Toothache (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 3 | 0
Chest pain (General disorders) | 2 | 0
Feeling cold (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Ulcer (General disorders) | 1 | 0
Hepatic pain (Hepatobiliary disorders) | 1 | 0
Hepatomegaly (Hepatobiliary disorders) | 3 | 0
Bronchitis (Infections and infestations) | 0 | 1
Otitis media chronic (Infections and infestations) | 0 | 1
Tuberculosis (Infections and infestations) | 1 | 3
Viral infection (Infections and infestations) | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 3
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0
Blood potassium increased (Investigations) | 1 | 0
Electrocardiogram ST-T change (Investigations) | 0 | 1
Reticulocyte count increased (Investigations) | 0 | 1
Weight decreased (Investigations) | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Intercostal neuralgia (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Alcoholism (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Hallucination (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 2 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 1 | 0
Peripheral coldness (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
The trial was terminated per protocol for lack of efficacy and not for dose limiting toxicity (DLT).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right to review results publications prior to public release and can delay such publications for a period greater than 60 days but no more than 120 days from the date that the publication is submitted to the Sponsor for review. Sponsor can require changes to the publication to protect Sponsor's intellectual property rights and/or confidential information and reserves the right to limit publication timing and scope of data published based on the number of study locations.